CLINICAL TRIAL: NCT03385681
Title: Pediatric Pain Management in Post Anesthesia Care Units - an Intervention Study
Brief Title: Pediatric Pain Management - an Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Nurses Organisation (Other); South-Eastern Norway Regional Health Authority (Other); London South Bank University (Other); Karolinska University Hospital (Other); Oslo Metropolitan University (Other); University of Oslo (Other); University Hospital, Akershus (Other); Helse Stavanger HF (Other Government); Haukeland University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Tone Rustøen, Senior Researcher, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014/7951; 2014/878 (Other: Regional Committee for Medical Research Ethics Norway)
Record Dates: First submitted 2017-10-30; First posted 2017-12-28 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Pain; Pediatric ALL
Keywords: pediatric pain; postoperative pain; pain assessment; pain management; knowledge; children; nurses
MeSH Terms: conditions — Pain, Postoperative; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Agnosia

STUDY DESIGN:
Intervention Model Description: Two parallell groups- intervention and control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The study will be conducted by nurses at 3 postoperative units with children and adolescents after surgery. All nurses working with patients in these units will be asked to participate. Tailored Educational Intervention is administered to this group.
  Interventions: Other: Tailored Educational Intervention
- Control Group (No Intervention): The study will be conducted by nurses at 3 postoperative units with children and adolescents after surgery. All nurses working with patients in these units will be asked to participate in the study.

INTERVENTIONS:
Other: Tailored Educational Intervention — The intervention will be a one-day seminar for nurses working at the units, with lectures and workshops with main focus on the subjects showing the lowest pediatric pain management competence. In addition, there will be clinical supervision in pediatric postoperative pain management (two or three days per unit). The intervention will be conducted by two experts (nurse and physician) in pediatric postoperative pain management. After the intervention there will be different reminders every week for the first month, and then every month (in different forms) about pediatric pain management during six months of time.
  Arms: Intervention Group

SUMMARY:
This study will explore nurses' pediatric postoperative pain management knowledge and clinical practices. The aim is to evaluate if a tailored educational intervention will improve nurses' knowledge and attitudes of pain management and pain management practices. The intervention offered is education and skills training. The study has a pre-post design and a comparison group. Data is collected before the intervention is started (baseline T1) and again one month (T2) and six months (T3) after the intervention. Nurses working in six postoperative units are participating. The units are the largest pediatric postoperative units of each of the six university hospitals covering all health regions in Norway. Three different approaches will be used to collect data (survey with questionnaire, observations of clinical practice, and interviews with children).

DETAILED DESCRIPTION:
The study will explore the nurses' pediatric postoperative pain management knowledge and clinical practice, and evaluate if a tailored educational intervention will improve postoperative pain management practice. This will be achieved by first exploring the pediatric postoperative pain management practice using different approaches (study 1). Then, an intervention will be developed based on the results from the first study and available research in the area (study 2). Finally, the investigators will investigate if the tailored interventions with nurses at postoperative units improve the nurses' knowledge of pediatric pain management (study 3).

Studies Activity:

Study 1: Explore nurses' pediatric postoperative pain practices.

Data collection (baseline T1):

* Knowledge and attitudes (questionnaire PNKAS-N)
* Observational study of nurses clinical practice
* Interview with children about pain and pain management after surgery

Study 2: Develop a tailored educational intervention

* Literature review
* Results from baseline
* Feedback from the head of the relevant units
* Staff views about the facilitators and barriers to optimized pediatric pain management

Study 3: Implementation and evaluation of the intervention

The intervention:

* Lectures and workshops for the included nurses
* Clinical supervision of the nurses

Data collection (one months after the intervention (T2), and six months after the intervention (T3))

* Questionnaire PNKAS-N (T2 and T3)
* Observational study of clinical practice (T2 and T3)
* Interview with children (T2)

ELIGIBILITY:
Inclusion Criteria:

Survey:

* nurses working in six postoperative units for children in six university hospitals in Norway

Observational study of clinical practice:

* nurses working in six postoperative units for children in six university hospitals in Norway
* children (0-18 years) and their parents admitted to these six postoperative units for children in six university hospitals in Norway during the data collection period

Interview with children:

* children older than six years going through surgery at the time of data collection at two of six units (randomly chosen), and their parents, will be asked to participate in this study

Exclusion Criteria:

Survey and Observational study of clinical practice:

* nurses not involved in clinical work
* nurses working part-time (less than 75%)

Interview with children:

* children not admitted to the postoperative units
* children younger than 6 years of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 876 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in nurses' knowledge and attitudes of pediatric pain management | short term - three months after baseline (one month after intervention) and long term - eight months after baseline (six months after intervention)
  Evaluated with "The Pediatric Nurses' Knowledge and Attitudes Survey Regarding Pain Questionnaire - Norwegian version" (PNKAS-N). Scale ranges from minimum 0 to maximum 40.

SECONDARY OUTCOMES:
Nurses pediatric pain management practices in postoperative units | baseline - after surgery (observing for two weeks in each unit)
  Evaluated with non-participant observation using a structured observational tool (checklist) and field notes
Changes in nurses' pediatric pain management practices in postoperative units | short term - three months after baseline (one month after intervention)
  Evaluated with non-participant observation using a structured observational tool (checklist) and field notes
Changes in nurses' pediatric pain management practices in postoperative units | long term - eight months after baseline (six months after intervention)
  Evaluated with non-participant observation using a structured observational tool (checklist) and field notes
Children's experiences of pain and pain management after surgery | baseline - after surgery
  Measured with Interview with children about postoperative pain using semi-structured interviews with children after surgery
Changes in children's experiences of pain and pain management after surgery | One month after intervention
  Evaluated with Interview with children about postoperative pain using semi-structured interviews with children after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tone Rustoen, PhD, Principal Investigator — Oslo University Hospital
Locations (6):
- Norway (6):
  - Haukeland University Hospital, Bergen
  - Akershus University hospital, Lillestrøm
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St. Olavs hospital Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT03385681/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT03385681/SAP_001.pdf